CLINICAL TRIAL: NCT05162339
Title: Inflammatory Bowel Disease and Thromboembolic Events
Status: Completed | Type: Observational
Sponsor: Centro Hospitalar Tondela-Viseu (Other)
Collaborators: Portuguese IBD Group (Unknown)
Responsible Party: Principal Investigator, Ana Carvalho, Principal Investigator, Centro Hospitalar Tondela-Viseu
Other Study IDs: CHTV07/2020.1
Record Dates: First submitted 2021-12-04; First posted 2021-12-17 (Actual); Last update posted 2021-12-17 (Actual); Status verified 2021-12

CONDITIONS: Inflammatory Bowel Diseases; Thromboembolism; Coagulation Disorder
MeSH Terms: conditions — Inflammatory Bowel Diseases; Thromboembolism; Hemostatic Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 36 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- IBD patients
  Interventions: Other: No intervention was made

INTERVENTIONS:
Other: No intervention was made — No intervention was made

SUMMARY:
The main objective was to demonstrate the existence and importance of hypercoagulability in patients with IBD, by determining the prevalence of changes in coagulation parameters and evaluating the impact of these changes on the occurrence of thromboembolic events.

ELIGIBILITY:
Inclusion Criteria:

* Patients with 18 years of age or older, diagnosed with IBD, followed at a gastroenterology consultation at Centro Hospitalar Tondela-Viseu, between November 2016 and April 2017.

Exclusion Criteria:

* Individuals with other risk factors for TE (severe hepatic or renal failure, valvular heart disease, atrial fibrillation, heart failure or cardiomyopathy, pregnancy, and oral anticoagulants or heparin at the baseline).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with 18 years of age or older, diagnosed with IBD (ECCO criteria), and followed at a gastroenterology consultation at Centro Hospitalar Tondela-Viseu
Sampling Method: Non-Probability Sample
Enrollment: 149 (Actual)
Dates: Start 2016-11-01 (Actual); Primary Completion 2020-04-30 (Actual); Study Completion 2020-04-30 (Actual)

PRIMARY OUTCOMES:
Prevalence of thromboembolic events in IBD | 36 months
  To evaluate the coagulation parameters and the prevalence of thromboembolic events in IBD patients
Coagulation parameters variations in IBD | 36 months
  To investigate the correlation between coagulation parameters and disease phenotype and activity.

CONTACTS AND LOCATIONS:
Locations (1):
- Centro Hospitalar Tondela Viseu, Viseu, Portugal

REFERENCES:
- [Derived] Carvalho AC, Pinho J, Cancela E, Vieira HM, Silva A, Ministro P. Inflammatory bowel disease and thromboembolic events: a c'lot to learn. Therap Adv Gastroenterol. 2022 May 25;15:17562848221100626. doi: 10.1177/17562848221100626. eCollection 2022. PMID 35651649